CLINICAL TRIAL: NCT04769284
Title: Psychological State of University Students of Health Sciences During COVID-19
Brief Title: Psychological State of Students of Health Sciences During COVID-19
Status: Completed | Type: Observational
Sponsor: Yolanda Marcen Roman (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Sponsor-Investigator, Yolanda Marcen Roman, Principal investigador, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Other Study IDs: Mental health student
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Stress, Psychological; Anxiety; Depression; Covid19
Keywords: university students; physical activity; gender stereotype
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression; COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mental health student — An ad-hoc questionnaire was designed that included sociodemographic variables related to the characteristics of the students. The variables sex, age, degree, employment situation, coexistence situation, economic situation, origin environment, country of origin, time of residence in the Spanish State were collected.
  Personal variables:
  * Gender stereotypes: Short version of the Bem Sex Rol Inventory (BRSI).
  * International Physical Activity Questionnaire (IPAQ)
  * Abbreviated Goldberg Anxiety Scale EADG
  * Modified version of EPP-10 related to COVID-19 (EPP-10-C)

SUMMARY:
University students report high levels of stress, anxiety and depression every year, which, according to some research, responsible for university administration and popular media, constitutes a global crisis of mental health of students at these levels.

Exposure to academic stress directly compromises students' motivation and attitudes towards learning.

High levels of perceived distress in the face of inadequate resources to deal with the situation leaves people at risk of developing major psychiatric problems, especially when this distress is prolonged or severe.

DETAILED DESCRIPTION:
Main goal:Study the impact of socio-demographic, personal and health factors that determine the performance / perception of pandemic stress) in students of Bachelor's degrees in Health Sciences.

Secondary objectives:

* Analyze the relationship between socio-demographic and personal characteristics and the perception of stress related to the Covid-19 pandemic.
* Identify the relationship between the perception of stress related to the Covid-19 pandemic and the role of gender / physical activity and the academic performance of undergraduate students in Health Sciences.

Methodology All variables will be obtained only once by means of a survey through google form. The questionnaire will be disseminated to all students of the degrees, by institutional email, through direct contact with the delegates of each course. After the first two weeks, a reminder will be made following the same routes. There will be no follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Students of the degree of nursing, occupational therapy and physiotherapy belonging to the Faculty of Health Sciences

Exclusion Criteria:

* Not belonging to any degree in Health Sciences of the Faculty of Health Sciences

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — men woman non-binary others
Study Population: The study population will be made up of nursing, physiotherapy and occupational therapy students from the Faculty of Health Sciences of Zaragoza. Students will be able to answer the questions through their electronic devices. At no time will it be known which student has responded since he is totally anonymous and voluntary.
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Modified version of EPP-10 related to COVID-19 (EPP-10-C) | 3 minutes
  EEP-10-C; modified version of the 10-item perceived stress scale (EEP-10), it is also composed of 10 items; each offers 5 response options: never, almost never, occasionally, almost always, and always. Items 1, 2, 3, 6, 9 and 10 are scored directly from 0 to 4 and items 4, 5, 7 and 8, conversely, from 4 to 0
Abbreviated Goldberg Anxiety Scale EADG | 3 minutes
  It examines four fundamental psychiatric areas: depression, anxiety, social inadequacy, and hypochondria. It contains 9 questions and the cut-off points are equal to or greater than 4 for the anxiety scale, and equal to or greater than 2 for the depression scale.

SECONDARY OUTCOMES:
Gender stereotypes: Short version of the Bem Sex Rol Inventory (BRSI). | 4 minutes
  The 12-item questionnaire collected 6 instrumental or masculine items (strong personality, acts as a leader, has the character of a leader, dominant personality, defender of their beliefs and makes decisions easily), and 6 expressive or feminine items (tender, gentle, warm, affectionate, understanding and sensitive to the needs of others). People answered each of the questions about their self-perception, using a 7-point Likert-type scale
Short International Physical Activity Questionnaire (IPAQ) | 4 minutes
  The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) carried out in the last seven days, as well as walking and sitting time in a work day.
  Reference Mets values are: walking 3.3 Mets, moderate physical activity: 4 Mets, vigorous physical activity: 8 Mets.

OTHER OUTCOMES:
Sociodemographic variables | 4 minutes
  An ad-hoc questionnaire was designed that included sociodemographic variables related to the characteristics of the students. The variables sex, age, qualification, employment situation, coexistence situation, economic situation, origin environment, country of origin were collected.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz F Rodríguez Roca, Study Director — Zaragoza´s University; Estela F Calatayud Sanz, Study Director — Zaragoza´s University; Isabel F Gómez Soria, Study Director — Zaragoza´s University; Ángel M Gasch Gallén, Study Director — Zaragoza´s University
Locations (1):
- Faculty of Health Sciences. Zaragoza's University, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The study design could be reported

REFERENCES:
- [Result] Bao Y, Sun Y, Meng S, Shi J, Lu L. 2019-nCoV epidemic: address mental health care to empower society. Lancet. 2020 Feb 22;395(10224):e37-e38. doi: 10.1016/S0140-6736(20)30309-3. Epub 2020 Feb 7. No abstract available. PMID 32043982
- [Result] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Result] Odriozola-Gonzalez P, Planchuelo-Gomez A, Irurtia MJ, de Luis-Garcia R. Psychological symptoms of the outbreak of the COVID-19 confinement in Spain. J Health Psychol. 2022 Mar;27(4):825-835. doi: 10.1177/1359105320967086. Epub 2020 Oct 30. PMID 33124471
- [Result] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Result] Adhikari SP, Meng S, Wu YJ, Mao YP, Ye RX, Wang QZ, Sun C, Sylvia S, Rozelle S, Raat H, Zhou H. Epidemiology, causes, clinical manifestation and diagnosis, prevention and control of coronavirus disease (COVID-19) during the early outbreak period: a scoping review. Infect Dis Poverty. 2020 Mar 17;9(1):29. doi: 10.1186/s40249-020-00646-x. PMID 32183901
- [Result] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Result] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789